CLINICAL TRIAL: NCT00999843
Title: Maintenance of Sorafenib Following Combined Therapy of Three-dimensional Conformal Radiation Therapy/Intensity-modulated Radiation Therapy and Transcatheter Arterial Chemoembolization in Patients With Locally Advanced Hepatocellular Carcinoma: a Phase I/II Study.
Brief Title: Safety Study of Sorafenib Following Combined Therapy of Radiation and TACE for Liver Cancer
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Guo-liang Jiang M.D., Fudan University Shanghai Cancer Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LCR-004
Record Dates: First submitted 2009-10-21; First posted 2009-10-22 (Estimated); Last update posted 2009-10-22 (Estimated); Status verified 2009-10

CONDITIONS: Hepatocellular Carcinoma
Keywords: Sorafenib; Three-dimensional conformal radiation therapy; Intensity-modulated radiation therapy; Transcatheter arterial chemoembolization
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Sorafenib — Sorafenib is administered only to the patients with non-progression disease (CR, PR and SD) 4 weeks after the completion of radiotherapy. The dose is 400 mg, p.o., twice a day. Sorafenib is continuously given for 12 months unless intolerable toxicities and/or tumor progression.

SUMMARY:
Patients with liver cancer will receive interventional therapy plus radiotherapy. Maintenance Sorafenib will be taken after the completion of radiotherapy. Hypothesis of the current study is that Sorafenib as a maintenance therapy is safe and superior to radiotherapy combined with interventional therapy in terms of survival in comparison to historical data.

DETAILED DESCRIPTION:
Patients with solitary lesion (bigger than 5 cm in diameter) histologically or cytologically confirmed HCC receive TACE (1-3 cycles) plus 3DCRT/IMRT 4-6 weeks later. Maintenance Sorafenib will be administered only for the patients with non-progression disease 4 to 6 weeks after the completion of radiotherapy. The dose will be 400 mg, p.o., twice a day. Sorafenib will be continuously given for 12 months unless intolerable toxicities and/or tumor progression. Hypothesis of the current study is that Sorafenib as a maintenance therapy after combined therapy of 3DCRT/IMRT and TACE is safe and superior to radiotherapy combined with TACE alone in terms of time to progression (TTP), progression-free survival (PFS) and overall survival (OS) in comparison to historical data.

ELIGIBILITY:
Inclusion Criteria:

1. Age of equal or older than 18 years and not over 75 years with a life expectancy of at least 12 weeks;
2. Karnofsky performance status (KPS) of ≥70;
3. Histologically or cytologically confirmed HCC;
4. BCLC stage B, solitary lesion (bigger than 5 cm in diameter) with tumor burden less than 50% of total liver volume;
5. Liver function of Child-Pugh A;
6. Technically unresectable, medically inoperable, or surgery declined by the patient;
7. Normal renal function and adequate bone marrow reservation;
8. Signed informed consent must be obtained prior to any study specific procedure.

Exclusion Criteria:

1. Presence of intrahepatic and/or extrahepatic metastases
2. Previous received systemic therapy for liver cancer;
3. History of radiotherapy to the liver;
4. Indistinct tumor boundary on CT/MRI images;
5. Previous or concurrent malignancies, with the exception of adequately treated basal cell carcinoma of the skin or in situ carcinoma of the cervix or superficial bladder tumors [Ta, Tis and T1];
6. History of cardiac disease: congestive heart failure > NYHA class 2, active CAD, cardiac arrythmias requiring anti-arrhythmic therapy or uncontrolled hypertension within the last 12 months;
7. Concurrent uncontrolled medical conditions;
8. Pregnancy or breast feeding;
9. Investigational drug therapy outside of this trial during or within 4 weeks of study entry;
10. Psychiatric or medical unstable conditions that compromise the patient's ability to give informed consent.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2009-10; Primary Completion 2010-10 (Estimated); Study Completion 2012-10 (Estimated)

PRIMARY OUTCOMES:
The safety and tolerability of maintenance Sorafenib. | twelve months

SECONDARY OUTCOMES:
Time to progression (TTP), progression-free survival (PFS) and overall survival (OS) | 30 months

CONTACTS AND LOCATIONS:
Overall Officials: Guo-liang Jiang, M.D., Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Zhao JD, Liu J, Ren ZG, Gu K, Zhou ZH, Li WT, Chen Z, Xu ZY, Liu LM, Jiang GL. Maintenance of Sorafenib following combined therapy of three-dimensional conformal radiation therapy/intensity-modulated radiation therapy and transcatheter arterial chemoembolization in patients with locally advanced hepatocellular carcinoma: a phase I/II study. Radiat Oncol. 2010 Feb 12;5:12. doi: 10.1186/1748-717X-5-12. PMID 20149262